CLINICAL TRIAL: NCT00114452
Title: A Phase 1 Randomized, Double-blind, Placebo-controlled, Dose Escalation, Multicenter Study to Determine the Safety of Intravenous Ex-vivo Cultured Adult Human Mesenchymal Stem Cells (Provacel) Following Acute Myocardial Infarction
Brief Title: Safety Study of Adult Mesenchymal Stem Cells (MSC) to Treat Acute Myocardial Infarction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mesoblast, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mesoblast, Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 401-402
Record Dates: First submitted 2005-06-14; First posted 2005-06-15 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Myocardial Infarction
Keywords: Acute Myocardial Infarction; Heart Attack; Cardiovascular Disease; Stem cells; Congestive Heart Failure; Heart Attack Repair
MeSH Terms: conditions — Myocardial Infarction; Cardiovascular Diseases; Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Provacel: Cohort 1 (Active Comparator): ex vivo cultured adult mesenchymal stem cells
  Interventions: Biological: Provacel
- Provacel: Cohort 2 (Active Comparator): ex vivo cultured adult mesenchymal stem cells
  Interventions: Biological: Provacel
- Provacel: Cohort 3 (Active Comparator): ex vivo cultured adult mesenchymal stem cells
  Interventions: Biological: Provacel
- Provacel: Cohort 4 (Active Comparator): ex vivo cultured adult mesenchymal stem cells
  Interventions: Biological: Provacel
- Placebo (Placebo Comparator): ex vivo cultured adult mesenchymal stem cells
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Provacel — ex vivo cultured adult mesenchymal stem cells
  Arms: Provacel: Cohort 1; Provacel: Cohort 2; Provacel: Cohort 3; Provacel: Cohort 4
Biological: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine whether adult stem cells [Provacel™(PUMP1)] are safe and possibly effective in the treatment of acute myocardial infarction (heart attack).

DETAILED DESCRIPTION:
Cardiovascular disease is the single largest killer of males and females in the United States with an average of 335,000 deaths per year. This year an estimated 700,000 Americans will suffer an acute myocardial infarction. The standard of care treatment for acute myocardial infarction (MI) usually includes immediate perfusion, optimal pain relief, oxygen, aspirin or other anti-coagulants, Beta-Blockers, nitrates and Ace-inhibitors. Management of cardiac risk factors such as tobacco use, hypertension, lipid levels, diabetes, weight control and exercise all work to reduce further atherosclerotic events. Yet, many patients go on to develop Congestive Heart Failure (CHF). Medical management for CHF may improve symptoms and slow the progression to failure but does not restore a functioning myocardium. A therapy that could improve the myocardial remodeling process and reduce the incidence or severity of CHF following acute MI would provide a significant benefit in an area of unmet medical need.

Patients will receive standard of care in addition to stem cells or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 21 and 85 years old
* First heart attack within 1 to 10 days

Exclusion Criteria:

* Positive for HIV 1 and 2
* Previous heart attack
* Pacemaker or other device
* Pregnant or breastfeeding
* Allergic to cow or pig derived products
* Previous bone marrow transplant
* Involved in another clinical trial within the past 30 days
* Alcohol or recreational drug abuse within the past 6 months
* Hepatitis Positive
* Major surgical procedure or major trauma within the past 14 days
* Body weight greater than 300 pounds
* Autoimmune disease ( e.g. Lupus, Multiple Sclerosis)

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-03-22 (Actual); Primary Completion 2006-10-04 (Actual); Study Completion 2008-04-24 (Actual)

PRIMARY OUTCOMES:
Comparison of treatment adverse event rates between the 0.5, 1.6 and 5.0 million mesenchymal stem cells per kilogram dose cohorts and placebo groups. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ken Borow, MD, Study Director — Mesoblast, Inc.
Locations (15):
- United States (15):
  - Arizona Heart Institute, Phoenix, Arizona
  - University of California - San Diego; Thornton, San Diego, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Rush University Medical Center, Chicago, Illinois
  - The Care Group, Indianapolis, Indiana
  - Jewish Hospital, Louisville, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Washington Adventist, Takoma Park, Maryland
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Columbia Presbyterian Hospital, New York, New York
  - University of Rochester - Strong Memorial, Rochester, New York
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Austin Heart Institute, Austin, Texas
  - Texas Medical School, Houston, Texas

REFERENCES:
- [Background] Orlic D, Hill JM, Arai AE. Stem cells for myocardial regeneration. Circ Res. 2002 Dec 13;91(12):1092-102. doi: 10.1161/01.res.0000046045.00846.b0. PMID 12480809
- [Background] Pittenger MF, Martin BJ. Mesenchymal stem cells and their potential as cardiac therapeutics. Circ Res. 2004 Jul 9;95(1):9-20. doi: 10.1161/01.RES.0000135902.99383.6f. PMID 15242981
- [Background] Shake JG, Gruber PJ, Baumgartner WA, Senechal G, Meyers J, Redmond JM, Pittenger MF, Martin BJ. Mesenchymal stem cell implantation in a swine myocardial infarct model: engraftment and functional effects. Ann Thorac Surg. 2002 Jun;73(6):1919-25; discussion 1926. doi: 10.1016/s0003-4975(02)03517-8. PMID 12078791
- [Derived] Hare JM, Traverse JH, Henry TD, Dib N, Strumpf RK, Schulman SP, Gerstenblith G, DeMaria AN, Denktas AE, Gammon RS, Hermiller JB Jr, Reisman MA, Schaer GL, Sherman W. A randomized, double-blind, placebo-controlled, dose-escalation study of intravenous adult human mesenchymal stem cells (prochymal) after acute myocardial infarction. J Am Coll Cardiol. 2009 Dec 8;54(24):2277-86. doi: 10.1016/j.jacc.2009.06.055. PMID 19958962
- See also: Click here for more information about heart disease — http://www.americanheart.org
- See also: Click here for more information about this study and adult mesenchymal stem cells. — http://www.osiris.com